CLINICAL TRIAL: NCT04032457
Title: PAVES Benchmarking Pilot Study of Daily Disposable Contact Lenses
Acronym: PAVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vision Service Plan (Industry)
Collaborators: Foresight Regulatory Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VS-19-01
Record Dates: First submitted 2019-04-17; First posted 2019-07-25 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Refractive Errors
Keywords: Contact Lens
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: Randomized cross-over after 1 week of wear of two lens brands.
Who Masked: Care Provider
Masking Description: Clinician masking achieved by clinic coordinator dispensing lenses. Open label to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (12):
- A1 - SiHyDD to Moist (Active Comparator): 1 week of Test SiHyDD contact lenses followed by cross over to 1 week of 1-DAY ACUVUE® Moist contact lenses.
  Interventions: Device: Phase A - olifilcon B with Tangible Coatings
- A2 - Moist to SiHyDD (Active Comparator): 1 week of 1-DAY ACUVUE® Moist contact lenses followed by cross over to 1 week of Test SiHyDD contact lenses.
  Interventions: Device: Phase A - olifilcon B with Tangible Coatings
- A3 - SiHyDD to OASDD (Active Comparator): 1 week of Test SiHyDD contact lenses followed by cross over to 1 week of ACUVUE® OASYS 1-Day contact lenses.
  Interventions: Device: Phase A - olifilcon B with Tangible Coatings
- A4 - OASDD to SiHyDD (Active Comparator): 1 week of ACUVUE® OASYS 1-Day contact lenses followed by cross over to 1 week of Test SiHyDD contact lenses.
  Interventions: Device: Phase A - olifilcon B with Tangible Coatings
- A5 - SiHyDD to DT1 (Active Comparator): 1 week of Test SiHyDD contact lenses followed by cross over to 1 week of Alcon DAILIES TOTAL 1® contact lenses.
  Interventions: Device: Phase A - olifilcon B with Tangible Coatings
- A6 - DT1 to SiHyDD (Active Comparator): 1 week of Alcon DAILIES TOTAL 1® contact lenses followed by cross over to 1 week of Test SiHyDD contact lenses.
  Interventions: Device: Phase A - olifilcon B with Tangible Coatings
- B1 - HydDD to Moist (Active Comparator): 1 week of Test HydDD contact lenses followed by cross over to 1 week of 1-DAY ACUVUE® Moist contact lenses.
  Interventions: Device: Phase B - etafilcon A with Tangible Coatings
- B2 - Moist to HydDD (Active Comparator): 1 week of 1-DAY ACUVUE® Moist contact lenses followed by cross over to 1 week of Test HydDD contact lenses.
  Interventions: Device: Phase B - etafilcon A with Tangible Coatings
- B3 - HydDD to BioTrue (Active Comparator): 1 week of Test HydDD contact lenses followed by cross over to 1 week of BIOTRUE ONEday® contact lenses.
  Interventions: Device: Phase B - etafilcon A with Tangible Coatings
- B4 - BioTrue to HydDD (Active Comparator): 1 week of BIOTRUE ONEday® contact lenses followed by cross over to 1 week of Test HydDD contact lenses.
  Interventions: Device: Phase B - etafilcon A with Tangible Coatings
- B5 - HydDD to AqCom+ (Active Comparator): 1 week of Test HydDD contact lenses followed by cross over to 1 week of DAILIES® AquaComfort PLUS® contact lenses.
  Interventions: Device: Phase B - etafilcon A with Tangible Coatings
- B6 - AqCom+ to HydDD (Active Comparator): 1 week of DAILIES® AquaComfort PLUS® contact lenses followed by cross over to 1 week of Test HydDD contact lenses.
  Interventions: Device: Phase B - etafilcon A with Tangible Coatings

INTERVENTIONS:
Device: Phase A - olifilcon B with Tangible Coatings — Daily disposable silicone hydrogel contact lens
  Arms: A1 - SiHyDD to Moist; A2 - Moist to SiHyDD; A3 - SiHyDD to OASDD; A4 - OASDD to SiHyDD; A5 - SiHyDD to DT1; A6 - DT1 to SiHyDD
Device: Phase B - etafilcon A with Tangible Coatings — Daily disposable hydrogel contact lens
  Arms: B1 - HydDD to Moist; B2 - Moist to HydDD; B3 - HydDD to BioTrue; B4 - BioTrue to HydDD; B5 - HydDD to AqCom+; B6 - AqCom+ to HydDD

SUMMARY:
The study will compare the short-term clinical performance and wearer and practitioner acceptability in a pilot study of a new-to-market spherical silicone hydrogel daily disposable soft contact lens (SiHyDD) to three (3) benchmark soft daily disposable lenses (DD) and, subsequently, of a new-to-market hydrogel spherical daily disposable (HydDD) soft contact lens to three (3) other hydrogel daily disposable lenses. .

The primary outcome variables for this study are subjective comfort and lens preference.

DETAILED DESCRIPTION:
The objective of the study is to compare the short-term clinical performance and wearer and practitioner acceptability in a pilot study of a new-to-market spherical silicone hydrogel olifilcon B with Tangible Coating daily disposable soft contact lens (SiHyDD) to three (3) benchmark soft daily disposable lenses (DD) and, subsequently, of a new-to-market hydrogel etafilcon A with Tangible Coating spherical daily disposable (HydDD) soft contact lens to three (3) other hydrogel daily disposable lenses. .

The primary outcome variables for this study are subjective comfort and lens preference.

ELIGIBILITY:
Inclusion Criteria:

* Healthy full-time wearers of spherical daily disposable contact lenses
* Vision correctable to 20/30 with spherical lenses in powers from +3.00 to +1.00 DS and from -1.00 to -7.00 DS
* Visual acuity corrected to at least 20/30 with spherical contact lens

Exclusion Criteria:

* Participating in another clinical trial
* Vision not correctable to 20/30 with lens powers listed above

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 144 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Subjective Lens Preference | Visit 3 - Approximately 2 weeks
  Subjective preference for either lens intervention or no preference. Likert question with forced preference for Test or Benchmark lens or no preference.

SECONDARY OUTCOMES:
8-item Contact Lens Dry Eye Questionnaire (CLDEQ-8) score | Visit 2 and 3 - Approximately 1 and 2 weeks, respectively
  Difference in CLDEQ-8 score with treatments relative to score with habitual lenses. The scale on the 8-item CLDEQ-8 instrument is from 1 to 33, with each item having a possible 4 or 5 points.

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Chalmers, OD, Principal Investigator — Clinical Trial Consultant
Locations (6):
- United States (6):
  - Ross Eyecare, Atlanta, Georgia
  - Professional Eye Care Center, Niles, Illinois
  - RevolutionEyes, Carmel, Indiana
  - Andover Optometry on Central, Andover, Massachusetts
  - Professional VisionCare, Westerville, Ohio
  - Primary Eyecare Group, PC, Brentwood, Tennessee

IPD SHARING:
Plan to Share IPD: No